CLINICAL TRIAL: NCT04743804
Title: A Phase 3, Randomized, Double-blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Ravulizumab in Adult Participants Who Have Thrombotic Microangiopathy Associated With a Trigger
Brief Title: Ravulizumab in Thrombotic Microangiopathy Associated With a Trigger
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment Challenges
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALXN1210-TMA-315; 2020-005328-13 (EudraCT Number)
Record Dates: First submitted 2021-01-28; First posted 2021-02-08 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Thrombotic Microangiopathy
Keywords: Complement; Trigger; Secondary thrombotic microangiopathy; Acute kidney injury
MeSH Terms: conditions — Thrombotic Microangiopathies; Acute Kidney Injury | interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ravulizumab (Experimental)
  Interventions: Biological: Ravulizumab; Other: Best Supportive Care
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo; Other: Best Supportive Care

INTERVENTIONS:
Biological: Ravulizumab — Body weight-based doses of ravulizumab will be administered intravenously as loading dose regimen followed by maintenance dosing every 8 weeks.
  Other Names: Ultomiris; ALXN1210
  Arms: Ravulizumab
Other: Placebo — Matching placebo
  Arms: Placebo
Other: Best Supportive Care — Participants will receive medications, therapies, and interventions per standard hospital treatment protocols (unless specifically prohibited by the protocol).

SUMMARY:
This study will investigate the efficacy and safety of ravulizumab compared to placebo in adult participants with thrombotic microangiopathy (TMA) associated with a trigger. Participants will be randomized to receive either ravulizumab plus best supportive care or placebo plus best supportive care. The treatment period is 26 weeks followed by a 26-week off-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Body weight ≥ 30 kilograms
3. Female participants of childbearing potential and male participants with female partners of childbearing potential must use highly effective contraception starting at screening and continuing until at least 8 months after the last dose of ravulizumab
4. TMA associated with a trigger (autoimmune disease, infection, solid organ transplant, drugs, and malignant hypertension)
5. Vaccinated against meningococcal infection (Neisseria meningitidis), within 3 years prior to, or at the time of, randomization. Participants who initiate study drug treatment less than 2 weeks after receiving a meningococcal vaccine must receive appropriate prophylactic antibiotics for at least 2 weeks after the vaccination. If participant cannot receive the meningococcal vaccine, then participant must be willing to receive antibiotic prophylaxis coverage against N. meningitidis during the entire Treatment Period and for 8 months following the final dose of study drug. Additional vaccination (Haemophilus influenzae type b (Hib) and Streptococcus pneumoniae) may be considered based on individual patient condition.

Exclusion Criteria:

1. Any known gene mutation that causes atypical hemolytic uremic syndrome (aHUS)
2. Postpartum aHUS
3. Known chronic kidney disease
4. TMA due to hematopoietic stem cell transplantation ≤ 12 months of Screening
5. Primary and secondary glomerular diseases other than lupus
6. Diagnosis of primary antiphospholipid antibody syndrome
7. Shiga toxin-producing Escherichia coli infections including but not limited to Shiga toxin-related hemolytic uremic syndrome
8. Known familial or acquired 'a disintegrin and metalloproteinase with a thrombospondin type 1 motif, member 13' (ADAMTS13) deficiency (activity < 5%)
9. Positive direct Coombs test which in the judgement of the Investigator is indicative of a clinically significant immune-mediated hemolysis not due to TMA
10. Clinical diagnosis of disseminated intravascular coagulation (DIC) in the judgement of the Investigator
11. Presence of sepsis requiring vasopressors within 7 days prior to or during Screening
12. Presence of monoclonal gammopathy including but not limited to multiple myeloma
13. Known bone marrow insufficiency or failure evidenced by cytopenias
14. Unresolved N. meningitidis infection
15. History of malignancy within 5 years of Screening with the exception of nonmelanoma skin cancer or carcinoma in situ of the cervix that has been treated with no evidence of recurrence
16. Use of any complement inhibitors within the past 3 years
17. Respiratory failure requiring mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (80):
- United States (17):
  - Research Site, Tucson, Arizona
  - Research Site, Orange, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, New York, New York
  - Research Site, Valhalla, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Salt Lake City, Utah
  - Research Site, Morgantown, West Virginia
- Belgium (5):
  - Research Site, Belgium
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (8):
  - Research Site, Belo Horizonte
  - Research Site, Botucatu
  - Research Site, Campinas
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (4):
  - Research Site, Kingston, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- France (6):
  - Research Site, Bordeaux
  - Research Site, Chambéry
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Tours
- Germany (2):
  - Research Site, Essen
  - Research Site, Hanover
- Italy (2):
  - Research Site, Bergamo
  - Research Site, Roma
- Japan (9):
  - Research Site, Bunkyō City
  - Research Site, Iruma-Gun
  - Research Site, Mitaka-shi
  - Research Site, Miyazaki
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Maastricht
  - Research Site, Nijmegen
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Gwangju
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
- United Kingdom (12):
  - Research Site, Bristol
  - Research Site, Carshalton
  - Research Site, Exeter
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Nottingham
  - Research Site, Oxford
  - Research Site, Salford
  - Research Site, Stevenage

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Werion A, Storms P, Zizi Y, Beguin C, Bernards J, Cambier JF, Dahan K, Dierickx D, Godefroid N, Hilbert P, Lambert C, Levtchenko E, Meyskens T, Poire X, van den Heuvel L, Claes KJ, Morelle J; UCLouvain TMA/HUS Network and KU Leuven TMA/HUS Network. Epidemiology, Outcomes, and Complement Gene Variants in Secondary Thrombotic Microangiopathies. Clin J Am Soc Nephrol. 2023 Jul 1;18(7):881-891. doi: 10.2215/CJN.0000000000000182. Epub 2023 Apr 21. PMID 37094330

RESULTS

PARTICIPANT FLOW:
Groups:
- Ravulizumab: Participants received weight-based dosages of ravulizumab for 26 weeks during the Initial Treatment Period. Participants received a loading dose of ravulizumab intravenously on Day 1, followed by maintenance dosing on Day 15 and once every 8 weeks thereafter.
- Placebo: Participants received weight-based dosages of placebo matched to ravulizumab for 26 weeks during the Initial Treatment Period. Participants received a loading dose of placebo matched to ravulizumab intravenously on Day 1, followed by maintenance dosing on Day 15 and once every 8 weeks thereafter.
Period: Overall Study
Arm/Group | Ravulizumab | Placebo
Started | 9 | 7
Received at Least 1 Dose of Study Drug | 9 | 7
Completed | 4 | 1
Not Completed | 5 | 6
Not completed — Other | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study Terminated by Sponsor | 1 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Death | 3 | 0

BASELINE CHARACTERISTICS:
Population: The Modified Intent-to-Treat Analysis Set included all randomized participants, excluding participants who enrolled prior to availability of ST-HUS and ADAMTS13 central laboratory results and were subsequently found to be ineligible after randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ravulizumab | Placebo | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (15.75) | 57.7 (17.70) | 52.4 (16.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Thrombotic Microangiopathy (TMA) Response at Week 26
Description: TMA response required the following: 1) Normalization of platelet count without transfusion support during the prior 7 days. 2) Normalization of LDH. 3) Improvement in glomerular filtration rate (eGFR) of >= 30% compared to baseline. Participants must meet each TMA criterion at 2 separate assessments obtained at least 24 hours apart, and any measurement in between.
Time Frame: Week 26
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 9 | 7
Participants | 2 | 3

2. Secondary Outcome: Time to Complete TMA Response
Description: The Kaplan-Meier estimate of time to event of complete TMA response is reported. TMA response required the following: 1) Normalization of platelet count without transfusion support during the prior 7 days. 2) Normalization of LDH. 3) Improvement in eGFR of >= 30% compared to baseline. Participants must meet each TMA criterion at 2 separate assessments obtained at least 24 hours apart, and any measurement in between. Participants who did not have a response were censored at the date of last visit or study discontinuation at the time when the analysis was performed.
Time Frame: Baseline through Week 26
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 2 | 3
days | NA [21.0 to NA] — Too few participants experienced the event to estimate the time to event median and upper limit of 95% CI. | NA [16.0 to NA] — Too few participants experienced the event to estimate the time to event median and upper limit of 95% CI.

3. Secondary Outcome: Number of Participants With Hematologic Response at Week 26
Description: Hematologic response required the following: (1) Normalization of platelet count without transfusion support during the prior 7 days, and (2) normalization of LDH.
Time Frame: Week 26
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 9 | 7
Participants | 5 | 6

4. Secondary Outcome: Number of Participants With Renal Response at Week 26
Description: Renal response is improvement in eGFR of >= 30% compared to baseline. If a participant is on dialysis ≤5 days prior to the date of eGFR assessment, the eGFR will be set to 10 milliliter/minute/1.73 meter square (mL/min/1.73 m^2) for that assessment. If a participant is on dialysis during the entire 26 week randomized Treatment Period, or through early discontinuation of study drug, then the change in eGFR was not calculated.
Time Frame: Week 26
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 9 | 7
Participants | 4 | 4

5. Secondary Outcome: Number of Participants On Dialysis at Week 26
Time Frame: Week 26
Population: The Modified Intent-to-Treat Analysis Set included all randomized participants, excluding participants who enrolled prior to availability of ST-HUS and ADAMTS13 central laboratory results and were subsequently found to be ineligible after randomization. Here, Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 5 | 4
Participants | 1 | 0

6. Secondary Outcome: Change From Baseline in eGFR at Week 26
Description: If a participant is on dialysis during the entire 26 week randomized Treatment Period, or through early discontinuation of study drug, then the change in eGFR was not calculated.
Time Frame: Baseline, Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliliter/minute/1.73 meter^2
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 5 | 4
milliliter/minute/1.73 meter^2 | 25.8 (19.90) | 17.5 (7.59)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 34
Description: The Safety Analysis Set included all participants who received at least 1 dose of study intervention.
Arm/Group | Ravulizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 3/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 6/9 | 3/7
Other Adverse Events (participants affected / at risk) | 9/9 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ravulizumab (N=9) | Placebo (N=7)
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Epstein-Barr viraemia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal pseudoaneurysm (Renal and urinary disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ravulizumab (N=9) | Placebo (N=7)
Nausea (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 3
Device related infection (Infections and infestations) | 1 | 1
Enterococcal infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Corynebacterium infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 2
Asthenia (General disorders) | 0 | 1
Catheter site pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Device related thrombosis (General disorders) | 0 | 1
Extravasation (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Illness (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Seizure (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Substance dependence (Psychiatric disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Oxygen saturation decreased (Investigations) | 2 | 0
Liver function test abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Cardiac contractility decreased (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Ventricular hypokinesia (Cardiac disorders) | 1 | 0
Drain site complication (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Euthyroid sick syndrome (Endocrine disorders) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Penile dermatitis (Reproductive system and breast disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to continued enrollment challenges, Alexion decided to terminate this study prematurely. There were no safety or efficacy concerns throughout the course of study. The planned interim analysis for sample size re-estimation and the planned primary analysis as specified in Protocol Amendment 2 were not conducted due to early termination of the study. No hypothesis testing or inferential statistical analysis for the purpose of treatment comparisons was performed due to small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT04743804/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT04743804/SAP_001.pdf